CLINICAL TRIAL: NCT05515692
Title: Pilot Study of Safety and Feasibility of Electron Beam Radiotherapy to Treat Refractory Sclerodermatous Chronic Graft-versus-Host Disease
Brief Title: Electron Beam Radiotherapy for the Treatment of Refractory Sclerodermatous Chronic Graft Versus Host Disease
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21382; NCI-2022-05914 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21382 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-08-17; First posted 2022-08-25 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm; Refractory Sclerodermatous Graft Versus Host Disease
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (electron beam radiotherapy) (Experimental): Patients undergo radiotherapy simulation on day -14 using either a clinical setup or CT simulation at the discretion of the treating radiation oncologist. Patients then undergo electron beam radiotherapy on day 0. Patients also undergo skin biopsies at baseline, day 28, and day 168 after radiotherapy, and high frequency ultrasound (HFUS) scans on days 28, 56, 84, 112, 140, and 168 after radiotherapy.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Combination Product: Electron Beam Therapy; Procedure: High Frequency Ultrasound Imaging; Other: Questionnaire Administration; Radiation: Radiation Therapy Treatment Planning and Simulation; Procedure: Skin Biopsy

INTERVENTIONS:
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo radiotherapy simulation using CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Combination Product: Electron Beam Therapy — Undergo electron beam radiotherapy
Procedure: High Frequency Ultrasound Imaging — Undergo HFUS
  Other Names: HFUS
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy Treatment Planning and Simulation — Undergo radiotherapy simulation using clinical setup
  Other Names: Radiation Therapy Treatment Planning/Simulation
Procedure: Skin Biopsy — Undergo biopsy
  Other Names: Biopsy of Skin

SUMMARY:
This clinical trial tests the safety and side effects of a single small dose (fraction) of electron beam radiotherapy (e-BRT) at 10 Gy dose in treating patients with refractory (did not respond to other treatments) sclerodermatous chronic graft versus host disease (GVHD). GVHD is the most common complication after bone marrow transplant from a donor and happens as a result of donor immune cells attacking patients cells. Fibroblasts are skin cells that produce collagen and fibers and are the cells mainly involved in development of skin GVHD. Previous research has shown that fibroblasts can become fibrocytes (inactive fibroblast) at the fastest rate after receiving 8 Gy or more radiation. Moreover, regulatory T cells (Tregs) are cells from the immune system that can control GVHD and previous research has shown that radiation can increase the number of Tregs. Therefore, e-BRT at 10 Gy has the potential to improve GVHD by increasing the fibroblast to fibrocyte speed and the number of Tregs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish safety of 10 Gy of 6 MeV electron beam radiotherapy (e-BRT) administration in subjects with refractory sclerodermatous chronic graft-versus-host disease (cGVHD).

SECONDARY OBJECTIVE:

I. To provide preliminary efficacy data on the anti-fibrotic effects of e-BRT treatment at 4 and 24 weeks.

EXPLORATORY OBJECTIVES:

I. To evaluate the skin microenvironment 21 days before (baseline) and 28, and 168 days after e-BRT administration by assessing the presence and percentage of immune cell subsets (including but not limited to Th17 and Treg cells), presence of fibroblast and fibrocytes, and changes in the vasculature as measured by microvessel density (MVD) by CD31 and VEGF staining in tissue microarrays (TMA).

II. To assess changes in the presence and levels of GVHD inflammatory biomarkers and cytokines (including but not limited to IL-17A, IL-21, and IL-2) in patients' plasma after treatment with e-BRT.

OUTLINE:

Patients undergo radiotherapy simulation on day -14 using either a clinical setup or computed tomography (CT) simulation at the discretion of the treating radiation oncologist. Patients then undergo electron beam radiotherapy on day 0. Patients also undergo skin biopsies at baseline, day 28, and day 168 after radiotherapy, and high frequency ultrasound (HFUS) scans on days 28, 56, 84, 112, 140, and 168 after radiotherapy.

After completion of the study, patients are followed up yearly.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Permitting to perform clinical photography
* Age: >= 18 years
* Histologically confirmed sclerodermatous GHVD
* Relapsed/refractory sclerodermatous cGVHD
* Measurable disease of at least 2.0 cm
* Failed at least >= 2 prior frontline therapies for sclerodermatous chronic GvHD
* Fully recovered from the acute toxic effects (except alopecia) to =< Grade 1 to prior therapy
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

  * To be performed within 7 days prior to Day 1 of protocol therapy unless otherwise stated
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 1 month after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Chemotherapy, radiation therapy, biological therapy, immunotherapy within 21 days prior to Day 1 of protocol therapy
* Herbal medications
* Females only: Pregnant or breastfeeding
* Inability to comprehend and sign inform consent
* Individuals known to carry germline gene mutations in TP53, NBS and ATM.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2024-09-18 (Estimated); Study Completion 2024-09-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity | From study initiation of study treatment to day 28
  Will be evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) version 5. Unacceptable toxicity (UT) is defined as any local toxicity at the level of the treatment portal that is greater or equal to Grade 3 per National Cancer Institute (NCI) CTCAE version 5.0. The observation window of UT is from receiving study treatment until day 28 or observation of UT, whichever comes first. Patients who receive study treatment and complete UT evaluation will be evaluable for UT. Patients who are inevaluable for UT will be replaced. Toxicity information recorded in each patient will include the type, severity, and the probable association with electron beam radiotherapy (eBRT). Tables will be constructed to summarize the observed incidence by severity and type of toxicity, and dose levels. All patients who receive eBRT will be included as part of an 'as treated' analysis, in toxicities/complications.

SECONDARY OUTCOMES:
Incidence of disease specific response | Up to day 168
  Disease-specific response criteria including, but not limited to: complete response (CR) and partial response (PR) according to the core clinician-assessed and patient-reported chronic graft versus host disease (GVHD)-specific measures recommended by National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-Versus-Host Disease: IV. The 2014 Response Criteria Working Group Report and modified Rodnan skin score, and 20 MHz ultrasound (US). The cumulative incidence of relapse/progression will be calculated as competing risks.
Incidence of disease specific response | Up to day 168
  Disease-specific response criteria including, but not limited to: complete response (CR) and partial response (PR) according to the core clinician-assessed and patient-reported chronic graft versus host disease (GVHD)-specific measures recommended by National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-Versus-Host Disease: IV. The 2014 Response Criteria Working Group Report and modified Rodnan skin score, and 20 MHz ultrasound (US). The cumulative incidence of non-relapse mortality will be calculated as competing risks.

CONTACTS AND LOCATIONS:
Overall Officials: Karamjeet S Sandhu, Principal Investigator — City of Hope Medical Center